CLINICAL TRIAL: NCT01913275
Title: Comparison Between Endoscopic Stenting and Cholecystojejunostomy for PreoperativeDrainage Before Pancreaticoduodenectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of interest
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peush Sahni, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIS/2/2001
Record Dates: First submitted 2011-05-10; First posted 2013-08-01 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Periampullary Cancer; Pancreatic Cancer
Keywords: cholecystojejunostomy; whipple's pancreaticoduodenectomy; endoscopic stenting; hyperbilirubinemia
MeSH Terms: conditions — Pancreatic Neoplasms; Hyperbilirubinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endoscopic stenting (Active Comparator): endoscopic stenting to reduce preoperative jaundice
  Interventions: Procedure: Endoscopic stenting
- cholecystojejunostomy (Active Comparator): surgical procedure to decrease preoperative jaundice
  Interventions: Procedure: cholecystojejunostomy

INTERVENTIONS:
Procedure: Endoscopic stenting — Endoscopic stenting to decrease preopertaive jaundice
  Arms: endoscopic stenting
Procedure: cholecystojejunostomy — surgical procedure to decrease preoperative jaundice
  Arms: cholecystojejunostomy

SUMMARY:
Periampullary carcinoma and carcinoma head of pancreas are common causes of obstruction at the lower end of the common bile duct. Whenever possible, surgical resection in the form of Whipple Pancreaticoduodenectomy (WPD) is the treatment of choice. However, this operation is associated with a substantial postoperative morbidity and mortality. With advances in surgical techniques and postoperative care there has been a decrease in the operative mortality. However, the postoperative morbidity remains high varying between 5%-64%. Of the various risk factors, the degree of jaundice as indicated by the serum bilirubin levels has been associated with an increased risk of complications. Preoperative biliary drainage has been tried to decrease the serum bilirubin levels and consequently decrease postoperative morbidity and mortality. Internal biliary drainage can be achieved by surgical cholecystojejunostomy or endoscopic bile duct stenting. Endoscopic stenting can be done as a day care procedure under conscious sedation, but involves insertion of a foreign body (stent), which results in introduction of bacteria into the bile and problems of postoperative infection. Also, endoscopic stenting before surgery may result in difficulty in dissecting around the common bile duct during the surgical procedure. While the surgical bilioenteric bypass has the advantage that no foreign body is inserted into the biliary tree and hence the likelihood of sepsis is low, it requires anesthesia and involves a surgical incision.

There is no study comparing the outcomes of preoperative endoscopic and surgical drainage in patients undergoing pancraticoduodenectomy. We plan to compare the outcomes of preoperative endoscopic biliary drainage with surgical drainage in patients undergoing pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Hypothesis preoperative biliary decompression by Cholecystojejunostomy will reduce infective complication by 23% as compared to endocopic stenting INTRODUCTION Pancreaticoduodenectomy has been associated with a substantial postoperative morbidity and mortality. Advances in surgical techniques and postoperative care have led to a decrease in the operative mortality. However, the postoperative morbidity has remained high varying between 5%-64%.1 Of the various risk factors, analyzed in the retrospective studies, the degree of jaundice as indicated by the serum bilirubin levels has been associated with an increased risk of complications.2-5 Preoperative biliary drainage has been tried to decrease the serum bilirubin levels and consequently decrease postoperative morbidity and mortality. However, its role remains controversial.

External biliary drainage using percutaneous transhepatic insertion of a catheter has been used.6,7 The disadvantages of external bleary drainage include the risk of spontaneous catheter dislodgement, inflammation and pain at the puncture site, leak of ascitic fluid and bile around the catheter, and loss of fluid and electrolytes. Moreover, bile has an antibacterial action and its loss has been associated with sepsis and renal failure. Hence, internal biliary drainage is considered more appropriate.

Internal biliary drainage can be achieved by surgical cholecystojejunostomy or endoscopic bile duct stenting. The internal drainage provides a more physiological route for drainage of bile into duodenum or jejunum, which prevents any loss of electrolytes and bile salts, and reduces the risk of endotoxemia. Two studies using endoscopic bilary drainage have shown benefit in terms of reduced postoperative morbidity and mortality.7,8 However, it involves the insertion of a foreign body (stent), which results in occurrence of bacteria in bile with its attendant problems of postoperative sepsis.

Prior to the availability of the endoscopic and percutaneous methods, surgical bilioenteric bypass was the only method for preoperative biliary decompression. The disadvantage of this method is that it requires anesthesia and involves a surgical incision. However, its advantages are that no foreign body is inserted into the biliary tree and hence the likelihood of sepsis is low. Also, endoscopic stenting before pancreaticoduodenectomy may result in difficulty while dissecting the common bile duct. Historically, Whipple conceived pancreaticoduodenectomy as a two staged procedure. The first stage was surgical decompression of biliary tract to reduce the level of the hyperbilirubinemia to minimize mortality and morbidity after extirepative surgery and the second stage was a definitive surgical resection.

There is no study comparing the outcomes of preoperative endoscopic and surgical drainage in patients undergoing pancraticoduodenectomy. We plan to carry out a randomized trial comparing the outcomes of preoperative endoscopic biliary drainage with surgical drainage in patients undergoing pancraticoduodenectomy.

AIMS AND OBJECTIVES

To compare endoscopic bilary stenting with cholecystojejunostomy as a preoperative biliary drainage procedure in patients undergoing pancreaticoduodenectomy with respect to

1. Technical success
2. Successful drainage
3. Procedural-related complications
4. Hospital stay
5. Intra-operative difficulty
6. Postoperative morbidity and mortality.

PATIENTS AND METHODS

All consecutive patients with surgical obstructive jaundice attending Gastrointestinal surgery and medicine OPD at AIIMS will be evaluated with a detailed history and clinical examination, liver function tests and an ultrasound abdomen. Those patients who have liver function tests and an ultrasound suggestive of lower end block will be further evaluated with a contrast enhanced CT and side viewing endoscopy (biopsy whenever possible) to characterize the nature of block.

Inclusion criteria

1. Patients with periampullary carcinoma and carcinoma of the head of pancreas.
2. Patients with serum bilirubin >15mg/dl

Exclusion criteria

1. Patients with gastric outlet obstruction.
2. Patients with unresectable tumour assessed by imaging techniques.
3. Patients with a history of cholecystectomy and Billroth II gastrectomy.
4. Patients stented outside Study design the number of patients to be included was calculated to be 67 in each group based on assumption that infective complications will be reduced to 7%. the sample size was calculated with power of 90% and alpha error of 0.5 Patients will be randomly divided using sealed envelope method (using computer generated random numbers) to two groups of 50patients each.

Group A: Endoscopic stenting Group B: Cholecystojejunostomy

Preprocedural preparation10

1. Informed consent: The patient will be explained about the course and nature of disease, alternatives methods of treatment available, outcome with and without treatment. The procedure will be explained completely to the patient including the risks and complications involved and then consent will be taken.
2. Investigations The following investigations will be done in all the patients

   1. Prothrombin time
   2. Liver function tests (LFTs)
   3. Baseline haematological, biochemical and radiological investigations done in all patients as follows:

   i) Haemogram ii) Kidney Function Test iii) Electrolytes iv) Blood sugar v) Chest X-ray vi) ECG
3. Prophylactic antibiotics: All patients will receive prophylactic antibiotics (Inj cefaperazone + sulbactam 1 gm) 2 hours before the procedure and these will be continued upto 72 hours after the procedure. Patients will be kept nil orally for 8 hours prior to the procedure, and will be well hydrated with i.v. fluids.

Procedure

1. Endoscopic stenting (EBS)11 A therapeutic duodenoscope and a standard sphincterotome will be used for canulation of the bile duct. A hydrophilic guidewire (Terumo, 0.032" dia or Jag wire 0.035" dia, microvasive) will be used to cross the malignant stricture. After the stricture was crossed with the help of a guidewire, the wire will be removed and bile will be aspirated. A small sphincterotomy will be done with a wire-guided sphincterotome to facilitate the passage of the stent. The sphincterotome will be removed and a guide catheter will be passed over the guidewire and then a 10 F 7 cm long straight plastic stent will be inserted across the stricture over the guidewire. A maximum of three attempts will be allowed for insertion of the stent after which it will be categorized as procedural failure.
2. Cholecystojejunostomy (CJ) Cholecystojejunostomy will be done under local anesthesia using a small subcostal incision made over the distended gall bladder. The anastomosis will be done in 2 layers using 3-0 vicryl and 3-0 silk sutures.

Any complications related to both procedures and following them will be recorded.

Follow up On day 5 following the endoscopic or surgical bypass, the patients will be reassessed clinically and with hematological and biochemical parameters with special reference to haemogram and LFTs to know whether the biliary drainage is effective. After 4 weeks along with clinical, hematological and biochemical parameters, nutritional parameters will also be assessed.

All patients will be considered for definitive procedure at least after 4 weeks after the biliary drainage procedure.

The operative difficulty, amount of blood loss, number of transfusions required and operative time during definitive surgery will be recorded. Following pancreaticoduodenectomy, the postoperative complications will be evaluated in both groups.

Outcome measures Primary

1. Technical success: Passage of a stent across the stricture, along with flow of bile through the stent.
2. Successful drainage: A decrease in bilirubin of at least 20% of the pretreatment value within 5 days after procedure
3. Procedure-related complication: was defined complications directly related to stent insertion/CJ
4. Intraoperative assessment: The operative difficulty, amount of blood loss, number of transfusions required and operative time during definitive surgery.

Secondary

1. Procedure-related mortality: was defined as death directly related to complications of stent insertion/CJ
2. Duration of hospital stay: Number of days in hospital from the time of surgery or stenting to initial discharge.
3. Postoperative complication: Complications occurring within 30 days after pancreaticoduodenectomy

   1. Wound infection: presence of purulent discharge with or without growth of microorganism or serous discharge that grows a pathogenic microorganism.
   2. Intra-abdominal abscess: when pus was drained, aspirated or discharged from the peritoneal cavity
   3. Postoperative haemorrhage: Hematemesis, malena, blood los from the abdominal wound or drian site requiring 2 or more units of blood transfusion.
   4. Pancreaticojejunal leak: Drain fluid amaylase level > 3 times the serum amylase on postoperative day 3 or beyond or percutaneous drainage of amylase rich intra-abdominal collection, with or without clinical sequelae such as fever, leucocytosis, fistula or abscess.
   5. Bile leak: Clinical bile leak or elevated bilirubin level in drain fluid with normal serum level.
4. Postoperative mortality: was defined as death within 30 days after surgery or before discharge from the hospital.

Stastistical analysis Baseline characteristic will be expressed in mean (SD). The Pearson chi square test and Fischer exact test will be used for to compare the categorical data as appropriate. The Student t-test will be used to compare the continuous variables. Multivariate analysis will be done using logistic regression tests. Length of hospital stay will be compared using the log-rank test and the Wilcoxon signed rank test. A pvalue of <0.05 will be taken as significant.

REFERENCES

1. Sastry RA, Sivam S. Routine preoperative biliary drainage of biliary tree must not be done in patients with obstructive jaundice. Debates in gastrointestinal surgery. Jabalpur- banarsidas Bhanot publishers. 1998:115-62
2. Povoski SP, Karpeh MS Jr, Conlon KC, Blumgart LH, Brennan MF. Association of preoperative biliary drainage with postoperative outcome following pancreaticoduodenectomy. Ann Surg 1999;230:131-42.
3. Grace PA, Pitt HA, Tompkins RK, DenBesten L, Longmire WP Jr. Decreased morbidity and mortality after pancreatoduodenectomy. Am J Surg 1986;151:141-9.
4. Kairaluoma MI, Stahlberg M, Kiviniemi H, Haukipuro K. Results of pancreatoduodenectomy for carcinoma of the head of the pancreas. Hepatogastroenterology 1989;36:412-8.
5. Blenkharn JI, Benjamin IS. Infection during percutaneous transhepatic biliary drainage. Surgery 1989;105:239.
6. Hatfield AR, Tobias R, Terblanche J, Girdwood AH, Fataar S, Harries-Jones R, et al. Preoperative external biliary drainage in obstructive jaundice. A prospective controlled clinical trial. Lancet 1982;23:896-9.
7. Denning DA, Ellison EC, Carey LC. Preoperative percutaneous transhepatic biliary decompression lowers operative morbidity in patients with obstructive jaundice. Am J Surg 1981;141:61-5.
8. Lygidakis NJ, van der Heyde MN, Lubbers MJ. Evaluation of preoperative biliary drainage in the surgical management of pancreatic head carcinoma. Acta Chir Scand 1987;153:665-8.
9. Whipple AO, Parson WB, Mullins LR. Treatment of carcinoma of ampulla of vater. Ann Surg 1935;102:763-9.
10. Gulati MS, Srinivasan A, Agarwal PP. Percutaneous Management of Malignant Biliary Obstruction: The Indian Perspective. Tropical Gastroenterology 2003;24:47-58.
11. Ahuja V, Garg PK, Kumar D, Goindi G, Tandon RK. Presence of white bile associated with lower survival in malignant biliary obstruction. Gastrointest Endosc 2002;55:186-91.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with periampullary carcinoma and carcinoma of the head of pancreas.
2. Patients with serum bilirubin >15mg/dl

Exclusion Criteria:

1. Patients with gastric outlet obstruction.
2. Patients with unresectable tumour assessed by imaging techniques.
3. Patients with a history of cholecystectomy and Billroth II gastrectomy.
4. Patients stented outside

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Technical success | 2 minutes
  Passage of a stent across the stricture, along with flow of bile through the stent
Successful drainage | 5 days
  A decrease in bilirubin of at least 20% of the pretreatment value within 5 days after procedure
Procedure-related complication: was defined complications directly related to stent insertion/CJ | 30 days
Intraoperative assessment | 0 hour
  The operative difficulty, amount of blood loss, number of transfusions required and operative time during definitive surgery.

SECONDARY OUTCOMES:
1. Procedure-related mortality | 30 days
  was defined as death directly related to complications of stent insertion/CJ
2. Duration of hospital stay | 30 days
  Number of days in hospital from the time of surgery or stenting to initial discharge.
3. Postoperative complication: | 30 days
  Complications occurring within 30 days after pancreaticoduodenectomy
a. Wound infection | 30 days
  presence of purulent discharge with or without growth of microorganism or serous discharge that grows a pathogenic microorganism.
b. Intra-abdominal abscess | 30 days
  when pus was drained, aspirated or discharged from the peritoneal cavity
c. Postoperative haemorrhage | 30 days
  Hematemesis, malena, blood los from the abdominal wound or drian site requiring 2 or more units of blood transfusion.
d. Pancreaticojejunal leak | 30 days
  Drain fluid amaylase level > 3 times the serum amylase on postoperative day 3 or beyond or percutaneous drainage of amylase rich intra-abdominal collection, with or without clinical sequelae such as fever, leucocytosis, fistula
e. Bile leak | 30 days
  Clinical bile leak or elevated bilirubin level in drain fluid with normal serum level.

CONTACTS AND LOCATIONS:
Overall Officials: Tushar K Chattopadhyay, MS, Study Director — Department of GI surgery All India Institute of medical sciences, New Delhi, India; Sundeep S Saluja, MCh, Principal Investigator — Department of GI surgery , All India Institute Of medical sciences, New Delhi, India
Locations (1):
- All India Institute of Medical sciences, New Delhi, India

REFERENCES:
- [Background] Povoski SP, Karpeh MS Jr, Conlon KC, Blumgart LH, Brennan MF. Association of preoperative biliary drainage with postoperative outcome following pancreaticoduodenectomy. Ann Surg. 1999 Aug;230(2):131-42. doi: 10.1097/00000658-199908000-00001. PMID 10450725